CLINICAL TRIAL: NCT00998933
Title: An Open-label Study of Serum Testosterone Levels in Non-dosed Females After Secondary Exposure to Testosterone Gel 1.62%
Brief Title: Study of Serum Testosterone Levels in Non-dosed Females After Secondary Exposure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Barbara Parker, Solvay Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S176.1.009
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Hypogonadism
Keywords: Testosterone replacement therapy
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Testosterone gel 1.62%

INTERVENTIONS:
Drug: Testosterone gel 1.62% — 5 grams applied topically to upper arms/shoulder and abdomen on Day 1

SUMMARY:
To further characterize the transfer potential of marketed testosterone gel and new 1.62% formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers, with a BMI 20-35 kg/m2 (males) and 20-30 kg/m2 (females).

Exclusion Criteria:

* Males: history, current or suspected prostate or breast cancer.
* Female: pregnant or lactating.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameters Total Testosterone AUC, Cav, Cmax | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (1):
- Site 1, Miami Gardens, Florida, United States

REFERENCES:
- [Derived] Stahlman J, Britto M, Fitzpatrick S, McWhirter C, Testino SA, Brennan JJ, Zumbrunnen TL. Serum testosterone levels in non-dosed females after secondary exposure to 1.62% testosterone gel: effects of clothing barrier on testosterone absorption. Curr Med Res Opin. 2012 Feb;28(2):291-301. doi: 10.1185/03007995.2011.652732. Epub 2012 Jan 24. PMID 22188558